CLINICAL TRIAL: NCT04273984
Title: Efficacy and Safety of Different Doses of Vaginal Misoprostol Prior to Intra Uterine Contraceptive Device Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, shiamaa ghazal helmy, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Misoprostol Prior to IUCD
Record Dates: First submitted 2020-02-10; First posted 2020-02-18 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Intra-uterine Device Complication
Keywords: misoprostol; IUCD
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1- Group 1 (misoprostol 200 mcg (Active Comparator): Group 1 :will take 1 tablet (200 mcg) of misoprostol and 1 placebo tablet,
  .,
  Interventions: Drug: Misoprostol
- 2- Group 2 (misoprostol 100 mcg) (Active Comparator): Group 2: will take1 tablet (100 mcg) of misoprostol and 1 placebo tablet,
  Interventions: Drug: Misoprostol
- 3- Group 3 (placebo group) (Placebo Comparator): Group 3 ): will take2 placebo tablets
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Tablets will be inserted digitally by an experienced gynecologist 3hours before IUD insertion with taking care not inserting the medication into the cervix.
  Other Names: misotac

SUMMARY:
investigators aim through this study to evaluate and compare the Safety and efficacy of different doses of misoprostol prior to IUCD insertion among women with nulliparous cervix beside the rate of occurrence of adverse effects.

DETAILED DESCRIPTION:
Today there is an ever-increasing variety of effective contraceptive methods. Although all have side effects, they offer a lower risk than that conferred by pregnancy Contraceptive methods are classified according to their effectiveness. The top tier offer the highest level of effectiveness (defined as <two pregnancies per 100 women per year) and fulfill the criteria of ease of use, long duration of action, minimal need for return visits to the clinic and minimal user motivation or intervention. These methods include intrauterine contraception, sub dermal contraceptive implants and male and female sterilization The American Congress of Obstetricians and Gynecologists encourages all women, especially adolescents, to use long-acting reversible contraception.

Although intrauterine devices (IUDs) are safe, reliable and highly effective forms of long- acting reversible contraception and has a very low failure rate (0.2-0.6 per 100 women per year) , it is used by only 7.6% and 14.5% of contraceptive users in developed and developing countries, respectively

According to the latest practice recommendations for contraceptive use by the Centers for Disease Control and Prevention, the potential barriers to IUD use include anticipated insertion pain and health care providers' concerns about difficult insertion ( It is therefore important to identify effective approaches to ease IUD insertion in order to overcome obstacles hindering IUD use

Insertion-associated pain is related to speculum insertion, tenaculum traction on the cervix, sounding of the uterus, passing of the insertion tube through the cervix and placement of the device within the uterine cavity

Failure of insertion occurs in up to 14% and 20% of parous and nulliparous women, respectively 13).

It has been suggested that difficulty and failure of insertion are experienced more in nulliparous women (adjusted odds ratio [AOR] 5.19; 95% confidence interval [CI] 2.49, 10.82) and in those with previous Caesarean delivery (AOR 5.38; 95% CI 2.58, 11.22), due to a narrower cervical os Fouda et al. found that women who had delivered only by Caesarean section experienced more pain with IUD insertion compared with women with previous vaginal delivery

Many investigators have studied how to minimize insertion pain or failure. Few studies, however, have assessed any measure to decrease pain or difficulty during IUD insertion in women with previous Caesarean delivery (and no prior vaginal delivery) Pergialiotis et al. conducted a meta-analysis of clinical trials of analgesic options for IUD placement. Owing to the small number of trials, however, they concluded that further studies were needed before a conclusion could be reached

Misoprostol is a synthetic analog of prostaglandin E1 originally approved for treatment and prevention of gastric ulcers induced by non steroidal anti inflammatory drugs. It can be administered sublingually, orally, vaginally, or rectally. Vaginal administration has been associated with the highest peak serum levels of misoprostol, and overall bioavailability is greatest for sublingual and vaginal administration.

Misoprostol has well-known cervical ripening and uterotonic effects, naturally leading to its use as an adjunct in many gynecologic procedures. Its use has been well studied in the hysteroscopy literature. Multiple well-designed studies have validated the efficacy of different doses of misoprostol before hysteroscopy in reducing pain with dilation, reducing the number of failed dilations, and increasing cervical canal diameter before dilation Given these data, it is reasonable to hypothesize that pretreatment with misoprostol could aid in IUD insertion.

As existing studies examining this question have asserted varied conclusions, through this study investigators will evaluate and compare the safety and efficacy of different doses of misoprostol prior to IUCD insertion among women with nulliparous cervix beside the rate of occurrence of adverse effects.

This study aims to compare the efficacy and safety of different doses of vaginal misoprostol prior to IUCD insertion among women with nulliparous cervix "those who never delivered vaginally".

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant,
* Nulliparous cervix: no previous vaginal delivery or any attempt of vaginal delivery,
* Seeking for IUD insertion,
* Signing an informed consent to participate in the study,

Exclusion Criteria:

* Pregnancy or signs of pregnancy,
* Signs of cervicitis,
* Any uterine abnormalities as congenital anomalies, endometrial lesions, adenomyosis, fibroids and intrauterine adhesions,
* Women with any kind of pelvic pain,
* Abnormal uterine bleeding,
* History of cervical surgery,• Vaginal delivery,
* Contraindication to misoprostol as allergy,
* Administration of any analgesics last 12h,
* Withdrawal of consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Pain scores | during insertion of IUCD
  Pain scores will be measured using a visual analogue scale (VAS) consisting of a 10 cm horizontal straight line on which 0 cm corresponded to no pain and 10 cm to the worst pain. The pain score will be measured within 5 min of insertion of the IUD tube.

SECONDARY OUTCOMES:
The ease of IUD insertion | during insertion ofIUCD
  The ease of IUD insertion: using the ease of insertion score (ES): a graduated VAS-like scale from 0 to 10; in which 10 means terribly difficult insertion and 0 means very easy insertion. The ES was validated for use in previous similar studies about IUD insertion (Abbas et al., 2017).
Successful IUD insertion | 5minutes after insertion of IUCD
  Successful IUD insertion which will be assessed by vaginal US device 'Samsung h 60' through the following criteria:
  * IUD is centrally located within the endometrial cavity
  * The crossbar is positioned in the fundal area.
  * The distance from the top of the uterine cavity to the IUD should be 3 mm or less. This ultrasound scan will be performed just after the IUCD insertion.
The duration of insertion in seconds | during insertion ofIUCD
  The duration of insertion in seconds: starting from putting loaded applicator at the external os till withdrawal of the applicator after IUD insertion
The women's level of satisfaction at the end of insertion | 1 miute after insertion of IUCD
  The women's level of satisfaction at the end of insertion: every woman will express her level of satisfaction with IUD insertion by completing a 10-cm VAS (with 0 = no satisfaction and 10
  = maximum satisfaction).

OTHER OUTCOMES:
The side effects of the study medication | within 3 hours from inserting the misoprostol tablet
  as shivering, nausea, vomiting and diarrhea
Complications from IUD insertion | during insertion ofIUCD
  as abdominal cramps, uterine bleeding, perforation and cervical trauma
The number of women who need additional analgesics after the insertion | 5 minutes after insertion
Failure of IUD insertion, due to technical difficulty or intolerance of the patient | during IUCD insertion

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed h Salama, MD.MRCOG, Study Director — Ainshams uinversity
Locations (2):
- Egypt (2):
  - Ain Shams University Maternity Hospital, Cairo
  - Misr University for Science & Technology, Cairo

REFERENCES:
- [Background] Abbas AM, Abdellah MS, Khalaf M, Bahloul M, Abdellah NH, Ali MK, Abdelmagied AM. Effect of cervical lidocaine-prilocaine cream on pain perception during copper T380A intrauterine device insertion among parous women: A randomized double-blind controlled trial. Contraception. 2017 Mar;95(3):251-256. doi: 10.1016/j.contraception.2016.10.011. Epub 2016 Nov 4. PMID 27823944
- [Background] Abdellah MS, Abbas AM, Hegazy AM, El-Nashar IM. Vaginal misoprostol prior to intrauterine device insertion in women delivered only by elective cesarean section: a randomized double-blind clinical trial. Contraception. 2017 Jun;95(6):538-543. doi: 10.1016/j.contraception.2017.01.003. Epub 2017 Jan 11. PMID 28088498
- [Background] Aronsson A, Fiala C, Stephansson O, Granath F, Watzer B, Schweer H, Gemzell-Danielsson K. Pharmacokinetic profiles up to 12 h after administration of vaginal, sublingual and slow-release oral misoprostol. Hum Reprod. 2007 Jul;22(7):1912-8. doi: 10.1093/humrep/dem098. Epub 2007 May 8. PMID 17488782
- [Background] Bahamondes MV, Espejo-Arce X, Bahamondes L. Effect of vaginal administration of misoprostol before intrauterine contraceptive insertion following previous insertion failure: a double blind RCT. Hum Reprod. 2015 Aug;30(8):1861-6. doi: 10.1093/humrep/dev137. Epub 2015 Jun 3. PMID 26040478